CLINICAL TRIAL: NCT06438705
Title: Clinical Application of a Novel 99mTc Labeled Fibroblast Activating Protein (FAP) Targeted Molecular Probe in Early Diagnosis of Tumors
Brief Title: 99mTc Labeled FAP Targeted Molecular Probe in Early Diagnosis of Tumors
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Feng Wang, Chief physician, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20240419-08
Record Dates: First submitted 2024-05-07; First posted 2024-06-03 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Tumor; Lung Cancer; Pancreatic Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: SPECT-CT imaging — The subjects were intravenously injected with 99mTc labeled FAPI imaging agent, and drank 300-500ml of water after administration. SPECT-CT imaging was performed 60 minutes later

SUMMARY:
At present, radiopharmaceuticals targeting FAP have been developed for the diagnosis and treatment of various tumors. Considering the problems of fast tumor tissue clearance and short retention time in small molecule FAP inhibitors based on quinoline rings, this project optimized their ligands and developed a new FAP targeted technetium labeled molecular imaging probe for SPECT/CT imaging research to evaluate its safety in clinical application and its effectiveness in tumor diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary subjects, patients or their legal representatives sign informed consent;
* Volunteers are of any gender and aged between 18 and 75 years old, including the cut-off value;
* Other imaging methods found tumor occupying;
* Patients with pre-treatment tumors for whom surgery or biopsy may be performed to obtain final pathological results.
* Kidney glomerular filtration rate(GFR)>50 ml/min, effective renal plasma flow(ERPF)>280 ml/min, platelet count (PLT) >75 000/μL, white blood cell (WBC) >3000/μL, alanine aminotransferase ALT, aspartate aminotransferase AST less than 3 times the normal value.

Exclusion Criteria:

* People who have a history of allergy to similar drugs , allergic constitution or are currently suffering from allergic diseases;
* Is conducting clinical research on other drugs, or has participated in clinical research on any drugs (excluding vitamins and minerals);
* Have other clinical problems that are difficult to control (such as hepatitis C virus infection or active hepatitis B, or other serious chronic infections and serious mental, neurological, cardiovascular, respiratory and other diseases);
* Obvious abnormal liver and kidney function, GFR less than 50 ml/min;
* Tumor load is greater than 50%, or there is obvious spinal cord compression;
* The expected survival period is less than half a year; Chemotherapy was performed within 6 months.
* Have severe acute concomitant diseases or serious refractory mental disorders;
* Pregnant and lactating women (where pregnancy is defined as a positive urine pregnancy study);
* Patients whose physical condition is not suitable for radiological examination;
* Other situations deemed inappropriate by the investigator to participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was mainly conducted by SPECT CT imaging, and a total of 20 cases were planned to be enrolled, which were evaluated by 2 attending physicians of nuclear medicine or above according to various measurement data of the subjects
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Tumor uptake | 1 hour after administering the probe
  Compare the lesion site with surrounding normal tissue to evaluate whether there is a significant increase in radioactive uptake. Select the lesion in the abnormal area of the image and draw a 3D area of interest (ROI) to obtain the average lesion volume count (T). Calculate the tumor target/non target value (T/NT) statistically

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No